CLINICAL TRIAL: NCT06536270
Title: Development of a Web-Based Food Frequency Questionnaire and Diet Quality Score for Turkish Adults: Validity and Reliability
Brief Title: Development of a Web-Based Food Frequency Questionnaire and Diet Quality Score for Turkish Adults
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Merve GÜNEY COŞKUN, Lecturer, Medipol University
Other Study IDs: E-10840098-772.02-6576
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Nutritional Assessments; Nutritional Quality
Keywords: Food Frequency Questionnaire; Dietary Assessment; Diet Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: A validation and reproducibility study with a cross-sectional component — The primary intervention in this study involves adapting and validating the eNutri web-based Food Frequency Questionnaire and Diet Quality Score for the Turkish population.

SUMMARY:
This research aims to adapt and validate the web-based eNutri Food Frequency Questionnaire (FFQ) and Diet Quality Score (DQS) for the Turkish population, addressing the current gap in dietary assessment tools for Turkey. The study involves adapting the UK-based eNutri FFQ to reflect Turkish dietary habits, including revising the food list, capturing portion size photos, and incorporating local food composition data. The revised FFQ will be validated against three 24-hour dietary recalls and tested for reproducibility.

DETAILED DESCRIPTION:
Background: Non-communicable diseases (NCDs), such as cardiovascular diseases, are important global health concerns. Accurate dietary assessment is pivotal in understanding the relationship between food intake and health outcomes. Presently, there is a notable absence of a comprehensive dietary assessment tool tailored for the Turkish population.

Objective: The primary objective of this research is to adapt and validate the web-based eNutri Food Frequency Questionnaire (FFQ) and Diet Quality Score (DQS) for the Turkish population, addressing the current gap in dietary assessment methods.

Design and Proposed Analysis: The first part of the study will involve adapting the UK-based e-Nutri FFQ to reflect dietary habits of Turkish adults (eNutri-Turkey), such as revising the food list, taking portion size photos, and incorporating Turkish food composition data. The revised FFQ delivered online will be validated against three 24-hour recalls by phone (reference method) and the FFQ will be administered twice to assess reproducibility. The study will employ Cronbach's Alpha for internal consistency and the Bland-Altman method for validity. Additionally, inter-rater reliability and reproducibility will be assessed through Cohen's Kappa and ICC analysis, respectively. The eNutri DQS will be adapted in accordance with Turkish dietary guidelines. Following the adaptation, its validity will be assessed using existing Turkish population nutrient data. This analysis will involve retrospectively calculating the DQS and examining its associations with key risk markers of chronic diseases (BMI, blood pressure, blood glucose and cholesterol levels). Additionally, two qualitative studies will be conducted before starting the validation study. Dietitians and nutrition academics from Turkey (n=10) will provide insights on the suitability and effectiveness of eNutri-Turkey through one-to-one interviews. Feedback received will be used to improve the FFQ and DQS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* No diagnosed medical conditions (e.g., diabetes, heart disease, cancer, gastrointestinal conditions).
* Not pregnant or lactating.
* No food allergies or intolerances.
* Not following a specialized diet (e.g., vegan, weight-loss, sports nutrition regimen; vegetarians are eligible).
* Not receiving face-to-face nutritional services or dietary advice from a medical professional.
* Not participating in another nutrition study.
* Residing in Turkey.

Exclusion Criteria:

* Individuals with any diagnosed medical conditions.
* Pregnant or lactating women.
* Individuals with food allergies or intolerances.
* Those following a specialized diet (except vegetarians).
* Participants currently receiving face-to-face nutritional services or dietary advice.
* Individuals involved in another nutrition study.
* Individuals residing outside of Turkey.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of Turkish adults aged 18-65 years who reside in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Validity of the web-based FFQ | 14-day period
  Assesses the validity of the adapted eNutri FFQ by comparing its results with those from three 24-hour dietary recalls. Validity is evaluated based on nutrient intake measurements.
Reproducibility of the web-based FFQ | 14-day period
  Measures reproducibility by administering the FFQ twice to participants and analyzing the consistency of the results. Consistency of results; statistical measures will be used for analysis.

SECONDARY OUTCOMES:
Usability of the web-based FFQ | Immediately after the first FFQ administration
  Evaluates usability through participant feedback on a scale (e.g., Likert scale) on the clarity and ease of use of the FFQ and portion size images.
Usability Comparison of 24-Hour Recall and web-based FFQ | Immediately after the second FFQ administration
  Compares dietary intake data obtained from the 24-hour recall method (reference method) with that obtained from the FFQ administered after the second FFQ to assess usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) sharing plan does not include making anonymized data available to other researchers. Instead, data access will be provided only through secure platforms to researchers with approved proposals, ensuring adherence to confidentiality and ethical standards. The data will be shared through publication, with clear terms outlined to safeguard participant privacy.